CLINICAL TRIAL: NCT05889676
Title: Validation of a Simultaneous Ocular/Cervical VEMP With Mastoid Vibration by B250
Acronym: BCVEMP By B250
Status: Active, not recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Luca Verrecchia, Principal investigator, Region Stockholm
Other Study IDs: K2023-3904
Record Dates: First submitted 2023-05-16; First posted 2023-06-05 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: VEMP by bone conduction — New bone conducted VEMP elicited by transducer B250

SUMMARY:
A Validation study in which the standard separate cVEMP and oVEMP will be compared with a new protocol in which the cVEMP and oVEMP can be recorded simultaneously in response to a mastoid vibration by bone transducer B250

ELIGIBILITY:
Inclusion Criteria:

-) dizzy patients attending the balance laboratory -

Exclusion Criteria:

-) age < 18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all adult patients attedning the balance laboratory at Karolinska University Hospital after written consent.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
response rate | during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Hearing and Balance Unit, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No